CLINICAL TRIAL: NCT07104071
Title: Effect of Light Brightness on Well-being, Breastfeeding Motivation, and Psychological Well-being of Postpartum Mothers: A Randomized Placebo-controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Yıldırım (Other)
Responsible Party: Sponsor-Investigator, Emine Yıldırım, Assistant professor, Osmaniye Korkut Ata University
Organization: Osmaniye Korkut Ata University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 131313
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Reduced Light Brightness
Keywords: peaces; well-being; breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): reduced light brightness
  Interventions: Other: reduced light brightness
- control group (No Intervention): No intervention

INTERVENTIONS:
Other: reduced light brightness — reduced light brightness
  Arms: Intervention group

SUMMARY:
This study aims to determine the effects of light brightness on postpartum mothers' well-being, breastfeeding motivation, and psychological well-being.

This study is a randomized, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* being postpartum mothers.

Exclusion Criteria:

* having communication problems

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-08-22 (Estimated); Study Completion 2025-08-23 (Estimated)

PRIMARY OUTCOMES:
peace scala | 12 hours
  peace
well-being scala | 12 hours
  well-being
breastfeeding motivation scala | 12 hours
  breastfeeding motivation

IPD SHARING:
Plan to Share IPD: No